CLINICAL TRIAL: NCT02475382
Title: Expanded Access Program With Nivolumab Monotherapy in Subjects With Advanced or Metastatic Squamous (Sq) or Non-Squamous (Non-Sq) Non-Small Cell Lung Cancer (NSCLC) Who Have Received at Least One Prior Systemic Regimens for the Treatment of Stage IIIb/IV SqNSCLC
Brief Title: Expanded Access Program With Nivolumab Therapy for Treatment of Advanced/Metastatic SqNSCLC or Non-SqNSCLC After One Prior Systemic Regimen
Acronym: CheckMate 169
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-169
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Squamous Non-Small Cell Lung Cancer; Non-squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days

SUMMARY:
The purpose of this study is to provide treatment with nivolumab, a fully human monoclonal antibody, to subjects who have relapsed after treatment with a minimum of 1 prior systemic treatment for advanced or metastatic squamous (Sq) or non-squamous (non-Sq) non-small cell lung cancer (NSCLC) , Stage IIIB/IV and whose physicians believe that nivolumab treatment is appropriate.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Sq or Non-Sq NSCLC, Stage IIIb/IV (histologically or cytologically confirmed)
* Relapsed after 1 prior platinum-based systemic treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
* CNS metastasis must be treated and returned to baseline at least 2 weeks before first dose of nivolumab and off steroids or using stable or decreasing dose of < 10 mg prednisone or equivalent
* Prior chemotherapy, Tyrosine Kinase Inhibitor (TKI) therapy or Immunotherapy (tumor vaccine, cytokine or growth factor to control cancer) must be completed at least 2 weeks before first nivolumab dose

Exclusion Criteria:

* CNS metastases (untreated and/or symptomatic)
* Carcinomatous meningitis
* ECOG Performance status > 3
* Corticosteroids > 10 mg prednisolone/day (or equivalent)
* Prior treatment with anti-PD-1, anti-PD-L-1, anti-PDL2, anti-CT137 or anti-CTLA antibody, including ipilimumab or any other drugs specifically targeting T cell costimulation or checkpoint pathways

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (37):
- Brazil (22):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Brasília, Federal District
  - Local Institution, Distrito Federal, Federal District
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Cascavel, Paraná
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Natal, Rio Grande do Norte
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Passo Fundo, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Florianópolis, Santa Catarina
  - Local Institution, Itajaí, Santa Catarina
  - Local Institution, Barretos, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, Ribeirão Preto, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, Salvador
  - Local Institution, São Paulo
- Canada (15):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Burnaby, British Columbia
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Richmond, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Chicoutimi, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Montreal, Quebec
  - Centre De Sante Et De Services Sociaux Rimouski Neigette, Rimouski, Quebec

REFERENCES:
- [Derived] Parodi D, Dighero E, Biddau G, D'Amico F, Bauckneht M, Marini C, Garbarino S, Campi C, Piana M, Sambuceti G. Localized FDG loss in lung cancer lesions. EJNMMI Res. 2024 Nov 1;14(1):102. doi: 10.1186/s13550-024-01161-y. PMID 39485534
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx